CLINICAL TRIAL: NCT04275206
Title: The Anti-inflammatory Effects of Harkány Medicinal Water
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pecs (Other)
Collaborators: National Research, Development and Innovation Office, Hungary (Unknown); Harkány Spa Hospital, Hungary (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 131531
Record Dates: First submitted 2020-02-14; First posted 2020-02-19 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Rheumatoid Arthritis; Psoriasis
Keywords: medicinal water,inflammation,biomarker,inflammatory disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Psoriasis

STUDY DESIGN:
Intervention Model Description: Psoriasis / RA (t=0) Control (t=1) ---> (t=3) Medicinal water (t=4) (t=0) Medicinal water (t=1) ---> (t=3) Control (t=4)
  After 6 months, treatments will be repeated, but transposed, the previously control patients will receive medicinal water treatment, and tap water treatment will be performed on the previously treated group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants: Tap water and medicinal water have the same pH, colour, smell; in another study we proved that they could not differentiate them.
  Care providers do not know if tap water or medicinal water was installed in the bath tub.
  Investigator: Control and treated patients are encoded. Outcome assessor can see only the encoded measurement results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medicinal water treated group (Experimental): 3-week-long inward rehabilitation, in a bath tab, for 30 min, 5 days a week. (After 6 months treatments will be repeated in tap water.)
  Interventions: Other: Harkány medicinal water
- Tap water treated group (Placebo Comparator): 3-week-long inward rehabilitation, in a bath tab, for 30 min, 5 days a week. (After 6 months treatments will be repeated in medicinal water.)
  Interventions: Other: Tap water (placebo control)

INTERVENTIONS:
Other: Harkány medicinal water — The aim is to prove the effectiveness of Harkány medicinal water on patients suffering from psoriasis and rheumatoid arthritis. The control group is treated with tap water.
  Arms: Medicinal water treated group
Other: Tap water (placebo control) — The control group is treated with tap water.
  Arms: Tap water treated group

SUMMARY:
The study aims to provide evidence on the effectiveness of Harkány medicinal water in psoriatic and rheumatoid arthritis patients using subjective and objective methods. It is a cross-over study, so first half of patients will receive medicinal water, the other half will receive tap water treatment, and after 6 months treatments will be repeated, but patients will receive the other type of water.

DETAILED DESCRIPTION:
Several studies have shown that medicinal waters are highly effective in the treatment of many diseases. Existing clinical trials were unable to provide scientific evidence by using the highest international standards to justify the efficiency of thermal waters. Harkány medicinal water has been used for rheumatic, skin and locomotor diseases for more than 100 years. Its beneficial effects are indisputable. However, to introduce these effects, internationally high-level scientific methods and investigations are needed.

Psoriasis is among the most common dermatological diseases worldwide. Its significance is emphasized by adverse effects on quality of life, caused by chronic pain, physical and psychical disability due to psoriatic plaques. Former studies revealed an increased risk of inflammatory bowel disease, cardiovascular disease and certain types of cancer. Moreover, excessive oxidative stress can be responsible for the onset of psoriasis complications.

Rheumatoid arthritis (RA) is an autoimmune disease responsible for significant morbidity, characterized by articular inflammation. Oxidative stress is a key marker for determining pathophysiology of patients with RA.

The pathophysiological link between these conditions is the presence of excessive oxidative stress.

Subjective methods will include questionnaires, objective markers of disease severity will include the measurement of biomarkers from blood samples.

ELIGIBILITY:
Inclusion Criteria:

* signed consent statement
* over 18 years of age
* lack of underlying renal disease (GFR >60 mL/min/1.73m2)
* lack of severe inflammation (WBC <20.000 G/l; CRP <50 mg/l; WE <40 mm/h)
* psoriasis vulgaris with skin lesions
* mild and inactive RA

Exclusion Criteria:

* having received any kind of balneotherapy within 1 year before admission
* discontinuance of rehabilitation
* withdrawal of consent
* clinically significant difference in severity of the patient's condition on 1st or 2nd admission
* severe RA
* patients suffering from cancer
* patients suffering from inflammatory bowel disease
* patients underwent stroke within 1 year
* severe hypercholesterolemia
* severe diabetes
* patients with renal insufficiency
* patients receiving any kind biological therapy
* patients whose medication has changed during the study period or one month prior to the second treatment session

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Dermatology Life Quality Index (DLQI) | baseline (on admission)
  Self reported questionnaire is to measure how much the skin problem has affected the patient's life over the last week.
  The scoring of each question is as follows:
  Very much - scored 3; A lot - scored 2; A little - scored 1; Not at all - scored 0; Not relevant - scored 0; Question 7, 'prevented work or studying' - scored 3.
  The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Functional Independence Measure (FIM) | baseline (on admission)
  It is an 18-item measurement tool that explores an individual's physical, psychological and social function. The tool is used to assess a patient's level of disability as well as change in patient status in response to rehabilitation or medical intervention.
  Each item is scored 1-7. No Helper: 7. Complete Independence (Timely, Safety); 6. Modified Independence (Device)
  Helper - Modified Dependence: 5. Supervision (Subject = 100%); 4. Minimal Assistance (Subject = 75% or more); 3. Moderate Assistance (Subject = 50% or more)
  Helper - Complete Dependence: 2. Maximal Assistance (Subject = 25% or more); 1. Total Assistance or not Testable (Subject less than 25%)
SF-36 | baseline (on admission)
  This questionnaire contains 36 items that assess patients' health status and its impact on their lives. SF-36 is a structured, self-report questionnaire that a patient can complete with little or no counseling from an interviewer. Answers to the questions yield eight domains [scored from 0 (low) to 100 (high)] and two summary physical and mental component scores (PCS and MCS).
Patient Uncertainty Questionnaire-Rheumatology (PUQ-R) | baseline (on admission)
  Questions about issues related to arthritis. Each item is scored 1-4 (1 = very uncertain, 4 = very certain). Patients answer each question according to how certain or uncertain they are about each issues.
Psoriasis Area Severity Index (PASI) | baseline (on admission)
  It is used to express the severity of psoriasis. It combines the severity (erythema, induration and desquamation) and percentage of affected area. For each body section (head, arms, trunk and legs) the percent of area of skin involved and the severity of three clinical signs (erythema, induration and desquamation) on a scale from 0 to 4 (from none to maximum) are to be specified.
Disease Activity Score Calculator for Rheumatoid Arthritis (DAS 28) | baseline (on admission)
  It makes an objective, reproducible and comparable assessment of the rheumatoid arthritis activity. It takes into account the following items:
  TJC28: The number of tender joints (0-28). SJC28: The number of swollen joints (0-28). ESR: The Erythrocyte Sedimentation Rate (in mm/h). GH: The patient global health assessment (from 0=best to 100=worst).
  The 28 tender or swollen joint scores target the same joints (shoulders, elbows, wrists, metacarpophalangeal joints, proximal interphalangeal joints and the knees).
White blood cell count (Routine laboratory parameter) | baseline (on admission)
  Aspecific test for monitoring inflammation.
Haemoglobin (Routine laboratory parameter) | baseline (on admission)
  Part of general laboratory test.
Haematocrit (Routine laboratory parameter) | baseline (on admission)
  Part of general laboratory test.
WE (Routine laboratory parameter) | baseline (on admission)
  Aspecific test for monitoring inflammation.
Creatinine /eGFR/ (Routine laboratory parameter) | baseline (on admission)
  General kidney function.
Uric acid (Routine laboratory parameter) | baseline (on admission)
  Aspecific marker of antioxidant system.
High sensitivity C-reactive protein (hs-CRP) | baseline (on admission)
  hs-CRP is an aspecific inflammatory parameter, involved in most risk evaluation systems and generally used in clinical practice.
Asymmetric dimethylarginine (ADMA) | baseline (on admission)
  ADMA is considered as a marker and mediator of oxidative stress and an indicator of vascular well-being.
Total antioxidant capacity (TAC) | baseline (on admission)
  TAC is an easily feasible, widely used method, indirect marker of oxidative stress.
Malondialdehyde (MDA) | baseline (on admission)
  MDA is a well-known biomarker of oxidative stress. It is also a sensitive marker of inflammation in patients with RA.

SECONDARY OUTCOMES:
Dermatology Life Quality Index (DLQI) | 3 weeks (before discharge)
  Self reported questionnaire is to measure how much the skin problem has affected the patient's life over the last week.
  The scoring of each question is as follows:
  Very much - scored 3; A lot - scored 2; A little - scored 1; Not at all - scored 0; Not relevant - scored 0; Question 7, 'prevented work or studying' - scored 3.
  The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Functional Independence Measure (FIM) | 3 weeks (before discharge)
  It is an 18-item measurement tool that explores an individual's physical, psychological and social function. The tool is used to assess a patient's level of disability as well as change in patient status in response to rehabilitation or medical intervention.
  Each item is scored 1-7. No Helper: 7. Complete Independence (Timely, Safety); 6. Modified Independence (Device)
  Helper - Modified Dependence: 5. Supervision (Subject = 100%); 4. Minimal Assistance (Subject = 75% or more); 3. Moderate Assistance (Subject = 50% or more)
  Helper - Complete Dependence: 2. Maximal Assistance (Subject = 25% or more); 1. Total Assistance or not Testable (Subject less than 25%)
SF-36 | 3 weeks (before discharge)
  This questionnaire contains 36 items that assess patients' health status and its impact on their lives. SF-36 is a structured, self-report questionnaire that a patient can complete with little or no counseling from an interviewer. Answers to the questions yield eight domains [scored from 0 (low) to 100 (high)] and two summary physical and mental component scores (PCS and MCS).
Patient Uncertainty Questionnaire-Rheumatology (PUQ-R) | 3 weeks (before discharge)
  Questions about issues related to arthritis. Each item is scored 1-4 (1 = very uncertain, 4 = very certain). Patients answer each question according to how certain or uncertain they are about each issues.
Psoriasis Area Severity Index (PASI) | 3 weeks (before discharge)
  It is used to express the severity of psoriasis. It combines the severity (erythema, induration and desquamation) and percentage of affected area. For each body section (head, arms, trunk and legs) the percent of area of skin involved and the severity of three clinical signs (erythema, induration and desquamation) on a scale from 0 to 4 (from none to maximum) are to be specified.
Disease Activity Score Calculator for Rheumatoid Arthritis (DAS 28) | 3 weeks (before discharge)
  It makes an objective, reproducible and comparable assessment of the rheumatoid arthritis activity. It takes into account the following items:
  TJC28: The number of tender joints (0-28). SJC28: The number of swollen joints (0-28). ESR: The Erythrocyte Sedimentation Rate (in mm/h). GH: The patient global health assessment (from 0=best to 100=worst).
  The 28 tender or swollen joint scores target the same joints (shoulders, elbows, wrists, metacarpophalangeal joints, proximal interphalangeal joints and the knees).
White blood cell count (Routine laboratory parameter) | 3 weeks (before discharge)
  Aspecific test for monitoring inflammation.
WE (Routine laboratory parameter) | 3 weeks (before discharge)
  Aspecific test for monitoring inflammation.
Creatinine /eGFR/ (Routine laboratory parameter) | 3 weeks (before discharge)
  General kidney function.
Uric acid (Routine laboratory parameter) | 3 weeks (before discharge)
  Aspecific marker of antioxidant system.
High sensitivity C-reactive protein (hs-CRP) | 3 weeks (before discharge)
  hs-CRP is an aspecific inflammatory parameter, involved in most risk evaluation systems and generally used in clinical practice.
Asymmetric dimethylarginine (ADMA) | 3 weeks (before discharge)
  ADMA is considered as a marker and mediator of oxidative stress and an indicator of vascular well-being.
Total antioxidant capacity (TAC) | 3 weeks (before discharge)
  TAC is an easily feasible, widely used method, indirect marker of oxidative stress.
Malondialdehyde (MDA) | 3 weeks (before discharge)
  MDA is a well-known biomarker of oxidative stress. It is also a sensitive marker of inflammation in patients with RA.

CONTACTS AND LOCATIONS:
Overall Officials: Katalin Dr Szendi, MD, PhD, Principal Investigator — University of Pecs
Locations (1):
- Katalin Dr Szendi, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 6 month of study completion.
Access Criteria: Requests will be reviewed and requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Szendi K, Gerencsér G, Murányi E, Varga Cs. Mutagenic activity of peloids in the Salmonella Ames test. Applied Clay Science 55: 70-74, 2012.
- [Background] Gerencsér G, Murányi E, Szendi K, Varga Cs. Ecotoxicological studies on Hungarian peloids (medicinal muds). Applied Clay Science 50(1): 47-50, 2010.
- [Background] Varga C, Laszlo M, Gerencser G, Gyongyi Z, Szendi K. Natural UV-protective organic matter in thermal water. J Photochem Photobiol B. 2015 Mar;144:8-10. doi: 10.1016/j.jphotobiol.2015.01.007. Epub 2015 Jan 22. PMID 25662041
- [Background] Gerencser G, Szendi K, Berenyi K, Varga C. Can the use of medical muds cause genotoxicity in eukaryotic cells? A trial using comet assay. Environ Geochem Health. 2015 Feb;37(1):63-70. doi: 10.1007/s10653-014-9630-7. Epub 2014 Jul 26. PMID 25063339
- [Background] Peter I, Jagicza A, Ajtay Z, Boncz I, Kiss I, Szendi K, Kustan P, Nemeth B. Balneotherapy in Psoriasis Rehabilitation. In Vivo. 2017 Nov-Dec;31(6):1163-1168. doi: 10.21873/invivo.11184. PMID 29102940
- [Background] Szendi K, Gyöngyi Z, Kontár Zs, Gerencsér G, Berényi K, Hanzel A, Fekete J, Kovács A, Varga Cs. Mutagenicity and Phthalate Level of Bottled Water Under Different Storage Conditions. Exposure and Health 10(1): 51-60, 2018.
- [Background] Hanzel A, Horvat K, Molics B, Berenyi K, Nemeth B, Szendi K, Varga C. Clinical improvement of patients with osteoarthritis using thermal mineral water at Szigetvar Spa-results of a randomised double-blind controlled study. Int J Biometeorol. 2018 Feb;62(2):253-259. doi: 10.1007/s00484-017-1446-6. Epub 2017 Sep 27. PMID 28956169
- [Background] Hanzel A, Berenyi K, Horvath K, Szendi K, Nemeth B, Varga C. Evidence for the therapeutic effect of the organic content in Szigetvar thermal water on osteoarthritis: a double-blind, randomized, controlled clinical trial. Int J Biometeorol. 2019 Apr;63(4):449-458. doi: 10.1007/s00484-019-01676-3. Epub 2019 Feb 7. PMID 30734126
- [Background] Nemeth B, Ajtay Z, Hejjel L, Ferenci T, Abram Z, Muranyi E, Kiss I. The issue of plasma asymmetric dimethylarginine reference range - A systematic review and meta-analysis. PLoS One. 2017 May 11;12(5):e0177493. doi: 10.1371/journal.pone.0177493. eCollection 2017. PMID 28494019
- [Background] Nemeth B, Kustan P, Nemeth A, Lenkey Z, Cziraki A, Kiss I, Sulyok E, Ajtay Z. [Asymmetric dimethylarginine: predictor of cardiovascular diseases?]. Orv Hetil. 2016 Mar 27;157(13):483-7. doi: 10.1556/650.2016.30396. Hungarian. PMID 26996894
- [Background] Peter I, Jagicza A, Ajtay Z, Kiss I, Nemeth B. [Psoriasis and oxidative stress]. Orv Hetil. 2016 Nov;157(45):1781-1785. doi: 10.1556/650.2016.30589. Hungarian. PMID 27817235
- [Background] Kalavacherla US, Ishaq M, Rao UR, Sachindranath A, Hepsiba T. Malondialdehyde as a sensitive marker of inflammation in patients with rheumatoid arthritis. J Assoc Physicians India. 1994 Oct;42(10):775-6. PMID 7876045